CLINICAL TRIAL: NCT03174002
Title: Handling Oxygenation Targets in Adults With Acute Hypoxaemic Respiratory Failure in the Intensive Care Unit: A Randomised Clinical Trial of a Lower Versus a Higher Oxygenation Target
Brief Title: Handling Oxygenation Targets in the Intensive Care Unit
Acronym: HOT-ICU
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other); Copenhagen Trial Unit, Center for Clinical Intervention Research (Other)
Responsible Party: Principal Investigator, Bodil Steen Rasmussen, Clinical Professor, MD, PhD, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AAUH-ICU-01; 2017-000632-34 (EudraCT Number)
Record Dates: First submitted 2017-05-30; First posted 2017-06-02 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Hypoxemic Respiratory Failure; Oxygen Toxicity
Keywords: Oxygenation; Acute Respiratory Distress Syndrome; Mechanical ventilation; Critical illness; Critical care
MeSH Terms: conditions — Respiratory Insufficiency; Respiratory Distress Syndrome; Critical Illness | interventions — Oxygen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low oxygenation target (Experimental): Partial pressure of oxygen in arterial blood (PaO2) 8 kPa (60 mmHg)
  Interventions: Drug: Oxygen
- High oxygenation target (Active Comparator): Partial pressure of oxygen in arterial blood (PaO2) 12 kPa (90 mmHg)
  Interventions: Drug: Oxygen

INTERVENTIONS:
Drug: Oxygen — Oxygen administration to achieve a PaO2 of 8 kPa (60 mmHg) from ICU admission to ICU discharge
  Other Names: Inspired oxygen
  Arms: Low oxygenation target
Drug: Oxygen — Oxygen administration to achieve a PaO2 of 12 kPa (90 mmHg) from ICU admission to ICU discharge
  Other Names: Inspired oxygen
  Arms: High oxygenation target

SUMMARY:
Handling oxygenation targets (HOT) is standard of care in the intensive care unit (ICU), however the quality and quantity of evidence is low and potential harm has been reported. The aim of the HOT-ICU trial is to assess the overall benefits and harms of two levels of oxygenation targets in adult critically ill patients with acute hypoxaemic respiratory failure in the ICU.

DETAILED DESCRIPTION:
Acutely ill adults with hypoxaemic respiratory failure admitted to the intensive care unit (ICU) are at risk of life-threatening hypoxia, and thus oxygen is administered. However, the evidence on the optimal level of oxygenation is of low quantity and quality with no firm evidence for benefit or harm. Importantly, liberal use of supplementary oxygen may increase the number of serious adverse events including death. The aim of the HOT-ICU trial is to assess the benefits and harms of two targets of partial pressure of oxygen in arterial blood (PaO2) in guiding the oxygen administration in acutely ill adults with hypoxaemic respiratory failure at ICU admission.

ELIGIBILITY:
Inclusion Criteria:

* Acutely admitted to the ICU AND
* Aged ≥ 18 years AND
* Receives supplemental oxygen with a flow of at least 10 L per minutes in an open system including high-flow systems OR at least a FiO2 of 0.50 in a closed system including invasive or non-invasive ventilation or CPAP systems AND
* Expected to receive supplemental oxygen for at least 24 hours in the ICU AND
* Having an arterial line for PaO2 monitoring

Exclusion Criteria:

* Cannot be randomised within twelve hours after present ICU admission
* Chronic mechanical ventilation for any reason
* Use of home oxygen
* Previous treatment with bleomycin
* Organ transplant during current hospital admission
* Withdrawal from active therapy or brain death deemed imminent
* Fertile woman (< 50 years of age) with positive urine human gonadotropin (hCG) or plasma-hCG
* Carbon monoxide poisoning
* Cyanide poisoning
* Methaemoglobinaemia
* Paraquat poisoning
* Any condition expected to involve the use of hyperbaric oxygen (HBO)
* Sickle cell disease
* Consent not obtainable according to national regulations
* Previously randomised into the HOT-ICU trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2928 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2020-11-03 (Actual); Study Completion 2021-08-03 (Actual)

PRIMARY OUTCOMES:
90-days mortality | 90 days
  Landmark mortality 90-days after randomisation

SECONDARY OUTCOMES:
Days alive without organ support | Within 90 days
  Percentage of days alive and free from mechanical ventilation, circulatory support and renal replacement therapy
Days alive out of the hospital | Within 90 days
  Percentage of days alive out of the hospital
Number of patients with one or more serious adverse events | Until ICU discharge, maximum 90 days
  Serious adverse events are defined as new episode of shock and new episodes of ischaemic events including myocardial or intestinal ischaemia or ischaemic stroke
1-year mortality | 1 year
  Landmark mortality 1 year after randomisation
Quality of life assessement using the EuroQual-5D-5L telephone interview in selcted sites | 1 year
  EQ-5D-5L 1-year after randomisation
Cognitive function 1-year after randomisation as assessed using the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) score in selected sites | 1 year
  RBANS score 1 year after randomisation at selected sites
Pulmonary function | 1 year
  Bodyplethysmography and carbon monooxide diffusion capacity 1 year after randomisation at sellected sites
A health economic analysis | 90 days
  The analytic details will be based on the result of the trial and specified (cost-effectiveness versus cost-minimisation analyses)

CONTACTS AND LOCATIONS:
Overall Officials: Bodil Steen Rasmussen, MD, PhD, Principal Investigator — Aalborg University Hospital, Denmark; Anders Perner, MD, PhD, Study Chair — Rigshospitalet, Denmark
Locations (37):
- Denmark (21):
  - Dept. of Intensive Care, Aalborg University Hospital, Aalborg
  - Dept. of Intensive Care East Section, Øst, Skejby, Aarhus University Hospital, Aarhus
  - Dept. of Intensive Care Section Nord, Skejby, Aarhus University Hospital, Aarhus
  - Dept. of Intensive Care, University Hospital Skejby, Aarhus
  - Dept. of Intensive Care 4131, Copenhagen University Hospital Rigshospitalet, Copenhagen
  - Dept. of Intensive Care, Bispebjerg Hospital, Copenhagen
  - Dept. of Intensive Care, Herlev Hospital, Herlev
  - Dept. of Intensive Care, Herning Hospital, Herning
  - Dept. of Intensive Care, Hillerød Hospital, Hillerød
  - Dept. of Intensive Care, Hjørring Hospital, Hjørring
  - Dept. of Intensive Care, Holbæk Hospital, Holbæk
  - Department of Intensive Care, Holstebro, Holstebro
  - Dept. of Intensive Care, Holstebro Hospital, Holstebro
  - Dept. of Intensive Care, Horsens Hospital, Horsens
  - Dept. of Intensive Care, Hvidovre Hospital, Hvidovre
  - Dept. of Intensive Care, Kolding Hospital, Kolding
  - Dept. of Intensive Care, Køge Hospital, Køge
  - Dept. of Intensive Care, Randers Hospital, Randers
  - Dept. of Intensive Care, Roskilde Hospital, Roskilde
  - Dept. of Intensive Care, Slagelse Hospital, Slagelse
  - Department of Intensive Care, Viborg Hospital, Viborg
- Finland (4):
  - Dept. of Intensive Care, Helsinki University Hospital, Helsinki
  - Dept. of Intensive Care, Central Finland Central Hospital, Jyväskylä
  - Dept. of Intensive Care, Kuopio University Hospital, Kuopio, Kuopio
  - Dept. of Intensive Care, Turku University Hospital, Turku, Turku
- Dept. of Intensive Care, Landspitali University Hospital Reykjavik, Reykjavik, Iceland
- Netherlands (2):
  - Dept. of Intensive Care, University Medical Center Groningen, Groningen
  - Dept. of Intensive Care, Canisius Wilhelmina Hospital, Nijmegen
- Dept. of Intensive Care, National Hospital, University of Oslo, Oslo, Norway
- Switzerland (2):
  - Dept. of Intensive Care, Basel University Hospital, Basel
  - Dept. of Intensive Care, Bern University Hospital, Bern
- United Kingdom (6):
  - Royal Berkshire NHS Foundation Trust, Reading, Berkshire
  - Department of Intensive Care, University Hospital of Wales, Cardiff, Wales
  - Kingston Hospital NHS Foundation Trust, Kingston upon Thames
  - Royal Glamorgan Hospital, Llantrisant
  - Manchester University NHS Foundation Trust, Manchester
  - Wythenshawe Hospital, Manchester

IPD SHARING:
Plan to Share IPD: Yes
All original records (incl. consent forms, eCRFs, and relevant correspondences) will be archived at trial sites for 15 years. The clean electronic trial database file will be delivered to the EudraCT Database and Zenodo (https://zenodo.org/about) and maintained for 15 years and anonymised if requested by the authorities.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Study Protocol and Statistical Analysis Plan has been published. Informed Consent Form are available on the webpage (www.cric.nu/hot-icu)
Access Criteria: Managed by the Steering Committee of the HOT-ICUT trial.
URL: https://www.cric.nu/hot-icu/

REFERENCES:
- [Background] Schjorring OL, Perner A, Wetterslev J, Lange T, Keus F, Laake JH, Okkonen M, Siegemund M, Morgan M, Thormar KM, Rasmussen BS; HOT-ICU Investigators. Handling Oxygenation Targets in the Intensive Care Unit (HOT-ICU)-Protocol for a randomised clinical trial comparing a lower vs a higher oxygenation target in adults with acute hypoxaemic respiratory failure. Acta Anaesthesiol Scand. 2019 Aug;63(7):956-965. doi: 10.1111/aas.13356. Epub 2019 Mar 18. PMID 30883686
- [Background] Barbateskovic M, Schjorring OL, Jakobsen JC, Meyhoff CS, Rasmussen BS, Perner A, Wetterslev J. Oxygen supplementation for critically ill patients-A protocol for a systematic review. Acta Anaesthesiol Scand. 2018 Aug;62(7):1020-1030. doi: 10.1111/aas.13127. Epub 2018 Apr 30. PMID 29708586
- [Background] Barbateskovic M, Schjorring OL, Russo Krauss S, Jakobsen JC, Meyhoff CS, Dahl RM, Rasmussen BS, Perner A, Wetterslev J. Higher versus lower fraction of inspired oxygen or targets of arterial oxygenation for adults admitted to the intensive care unit. Cochrane Database Syst Rev. 2019 Nov 27;2019(11):CD012631. doi: 10.1002/14651858.CD012631.pub2. PMID 31773728
- [Background] Rasmussen BS, Perner A, Wetterslev J, Meyhoff CS, Schjorring OL. Oxygenation targets in acutely ill patients: still a matter of debate. Lancet. 2018 Dec 8;392(10163):2436-2437. doi: 10.1016/S0140-6736(18)32201-3. No abstract available. PMID 30527413
- [Background] Schjorring OL, Klitgaard TL, Perner A, Wetterslev J, Lange T, Keus F, Laake JH, Morgan M, Backlund M, Siegemund M, Thormar KM, Rasmussen BS. The handling oxygenation targets in the intensive care unit (HOT-ICU) trial: Detailed statistical analysis plan. Acta Anaesthesiol Scand. 2020 Jul;64(6):847-856. doi: 10.1111/aas.13569. Epub 2020 Mar 4. PMID 32068884
- [Derived] Nielsen MB, Klitgaard TL, Weinreich UM, Nielsen FM, Perner A, Schjorring OL, Rasmussen BS. Effects of a lower versus a higher oxygenation target in intensive care unit patients with chronic obstructive pulmonary disease and acute hypoxaemic respiratory failure: a subgroup analysis of a randomised clinical trial. BJA Open. 2024 Apr 29;10:100281. doi: 10.1016/j.bjao.2024.100281. eCollection 2024 Jun. PMID 38711834
- [Derived] Klitgaard TL, Schjorring OL, Severinsen MT, Perner A, Rasmussen BS. Lower versus higher oxygenation targets in ICU patients with haematological malignancy - insights from the HOT-ICU trial. BJA Open. 2022 Sep 23;4:100090. doi: 10.1016/j.bjao.2022.100090. eCollection 2022 Dec. PMID 37588787
- [Derived] Crescioli E, Lass Klitgaard T, Perner A, Lilleholt Schjorring O, Steen Rasmussen B. Lower versus higher oxygenation targets in hypoxaemic ICU patients after cardiac arrest. Resuscitation. 2023 Jul;188:109838. doi: 10.1016/j.resuscitation.2023.109838. Epub 2023 May 16. PMID 37196799
- [Derived] Crescioli E, Klitgaard TL, Poulsen LM, Brand BA, Siegemund M, Grofte T, Keus F, Pedersen UG, Backlund M, Karttunen J, Morgan M, Ciubotariu A, Bunzel AG, Vestergaard SR, Jensen NM, Jensen TS, Kjaer MN, Jensen AKG, Lange T, Wetterslev J, Perner A, Schjorring OL, Rasmussen BS. Long-term mortality and health-related quality of life of lower versus higher oxygenation targets in ICU patients with severe hypoxaemia. Intensive Care Med. 2022 Jun;48(6):714-722. doi: 10.1007/s00134-022-06695-0. Epub 2022 Apr 20. PMID 35441849
- [Derived] Klitgaard TL, Schjorring OL, Lange T, Moller MH, Perner A, Rasmussen BS, Granholm A. Lower versus higher oxygenation targets in critically ill patients with severe hypoxaemia: secondary Bayesian analysis to explore heterogeneous treatment effects in the Handling Oxygenation Targets in the Intensive Care Unit (HOT-ICU) trial. Br J Anaesth. 2022 Jan;128(1):55-64. doi: 10.1016/j.bja.2021.09.010. Epub 2021 Oct 19. PMID 34674834
- [Derived] Rasmussen BS, Klitgaard TL, Perner A, Brand BA, Hildebrandt T, Siegemund M, Hollinger A, Aagaard SR, Bestle MH, Marcussen KV, Brochner AC, Solling CG, Poulsen LM, Laake JH, Aslam TN, Backlund M, Okkonen M, Morgan M, Sharman M, Lange T, Wetterslev J, Schjorring OL. Oxygenation targets in ICU patients with COVID-19: A post hoc subgroup analysis of the HOT-ICU trial. Acta Anaesthesiol Scand. 2022 Jan;66(1):76-84. doi: 10.1111/aas.13977. Epub 2021 Sep 20. PMID 34425016
- [Derived] Schjorring OL, Klitgaard TL, Perner A, Wetterslev J, Lange T, Siegemund M, Backlund M, Keus F, Laake JH, Morgan M, Thormar KM, Rosborg SA, Bisgaard J, Erntgaard AES, Lynnerup AH, Pedersen RL, Crescioli E, Gielstrup TC, Behzadi MT, Poulsen LM, Estrup S, Laigaard JP, Andersen C, Mortensen CB, Brand BA, White J, Jarnvig IL, Moller MH, Quist L, Bestle MH, Schonemann-Lund M, Kamper MK, Hindborg M, Hollinger A, Gebhard CE, Zellweger N, Meyhoff CS, Hjort M, Bech LK, Grofte T, Bundgaard H, Ostergaard LHM, Thyo MA, Hildebrandt T, Uslu B, Solling CG, Moller-Nielsen N, Brochner AC, Borup M, Okkonen M, Dieperink W, Pedersen UG, Andreasen AS, Buus L, Aslam TN, Winding RR, Schefold JC, Thorup SB, Iversen SA, Engstrom J, Kjaer MN, Rasmussen BS; HOT-ICU Investigators. Lower or Higher Oxygenation Targets for Acute Hypoxemic Respiratory Failure. N Engl J Med. 2021 Apr 8;384(14):1301-1311. doi: 10.1056/NEJMoa2032510. Epub 2021 Jan 20. PMID 33471452
- [Derived] Klitgaard TL, Schjorring OL, Lange T, Moller MH, Perner A, Rasmussen BS, Granholm A. Bayesian and heterogeneity of treatment effect analyses of the HOT-ICU trial-A secondary analysis protocol. Acta Anaesthesiol Scand. 2020 Oct;64(9):1376-1381. doi: 10.1111/aas.13669. Epub 2020 Aug 5. PMID 32659856
- See also: Link to the HOT-ICU website — https://www.cric.nu/hot-icu/